CLINICAL TRIAL: NCT05224570
Title: Epidemiology of Gunshot Wounds Injuries Admitted in Intensive Care Unit in France: a Retrospective Multicenter Observational Study
Brief Title: Epidemiology of Gunshot Wounds Injuries Admitted in ICU in France
Acronym: GSW_in_ICU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/LR-01
Record Dates: First submitted 2021-08-16; First posted 2022-02-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2022-01

CONDITIONS: Gunshot Wound
MeSH Terms: conditions — Wounds, Gunshot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gunshot wounds admitted in ICU: patient with Gunshot wounds admitted to ICU

SUMMARY:
In civilian practice, the incidence of firearm violence depends on the country. In high income countries, most cases are reported in the USA or South Africa. In these countries, gunshot wounds (GSW) represent 20% of death cases in trauma centers, more than motor vehicle collisions.

The mortality in civilian practice occurs during the first 24 hours following GSW, mainly due to hemorrhage and traumatic brain injury, though long term effects on physical and psychological outcomes have also been shown.

Some factors of mortality specific to GSW have been established: multiples wounds, homicide vs suicide attempt, impact zone, or firearm caliber.

Few specific guidelines have been published concerning civilian GSW management. These cases are mostly treated in standard guidelines, such as hemorrhagic shock or traumatic brain injury guidelines. As in other trauma mechanisms, the "platinum ten minutes and golden hour" concept is applicable.

In Europe, the incidence of civilian GSW is much lower and few European studies have been published recently. Penetrating injuries in Europe are less likely to be GSW, and are more often self-inflicted than in the USA. In addition, European studies are heterogeneous, due to the difference in populations, healthcare systems and GSW being grouped with stabbing wounds under the label "penetrating trauma".

However, there is a global concern in Europe regarding a potential rise of GSW, with higher severity score than conventional trauma patients and often necessitate ICU admission. Studies analyzing data from different European countries show significantly different ICU admission rates for overall GSW, ranging from 17% up to 30%.

Therefore, the investigators conducted a multicenter, retrospective study on four French University Hospitals aiming to describe the epidemiology (mortality and type of organ damage) and identify prognosis factors of civilian GSW admitted in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Admission for gunshot wound care in ICU between 1st of January 2015 and June 30th 2021 at Nimes University Hospital, Marseille North University Hospital, Montpellier University Hospital, Toulon Military Teaching Hospital.
* Patient ≥ 15 years old

Exclusion Criteria:

* Patient < 15 years old
* Patient who objected to the use of their data.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who were admitted for gunshot wound care in ICU between 1st of January 2015 and June 30th 2021 at Nîmes University Hospital, Marseille North University Hospital, Montpellier DAR_A University Hospital, Toulon Military Teaching Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Mortality | day 28
  mortality rate at day 28 of patients admitted for Gunshot wounds

SECONDARY OUTCOMES:
Age | Day 0
  To identify if age is a prognosis factors of mortality of patients admitted for Gunshot
Sex | Day 0
  To identify if sex is a prognosis factors of mortality of patients admitted for Gunshot
Comorbidity | Day 0
  To identify if some comorbidities are some prognosis factors of mortality of patients admitted for Gunshot wounds (age, sex, comorbidity, type of gunshot, bullet impact zone, delay to reach hospital, biological parameters at ICU admission, use of antibiotics, blood transfusion, type of surgery, medical management, initiation of renal replacement therapy, length of ICU stay, ).
Type of gunshot | Day 0
  To identify if the type of gunshot is prognosis factors of mortality of patients admitted for Gunshot wounds
Bullet impact zone | Day 0
  To identify if the impact zone is a prognosis factors of mortality of patients admitted for Gunshot wounds
Delay to reach hospital | Day 0
  To identify if the delay to reach hospital is a prognosis factors of mortality of patients admitted for Gunshot wounds
biological parameters at ICU admission | Day 0
  To identify if some biological parameters at admission are prognosis factors of mortality of patients admitted for Gunshot wounds
antibiotics cure | Day 0
  To identify if an antibiotic cure at admission is a prognosis factors of mortality of patients admitted for Gunshot wounds
Blood transfusion | Day 0 to day 30
  To identify if a blood transfusion is a prognosis factors of mortality of patients admitted for Gunshot wounds
Type of surgery | Day 0 to day 30
  To identify if surgery type is a prognosis factors of mortality of patients admitted for Gunshot wounds
renal replacement therapy | Day 0 to day 30
  To identify if initiation of renal replacement therapy is a prognosis factors of mortality of patients admitted for Gunshot wounds
length of ICU stay | Day 0 to day 30
  To identify if length of ICU stay is a prognosis factors of mortality of patients admitted for Gunshot wounds

CONTACTS AND LOCATIONS:
Overall Officials: Loic ROUGERIE, Principal Investigator — CHU NIMES; Laurent MULLER, Md, PhD, Study Director — CHU NIMES
Locations (1):
- CHU de NIMES, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rougerie L, Charbit J, Mezzarobba M, Leone M, Duclos G, Meaudre E, Cungi PJ, Bartoli C, Thierry GR, Roger C, Muller L. Epidemiology of civilian's gunshot wound injuries admitted to intensive care unit: A retrospective, multi-center study. Injury. 2024 Oct;55(10):111735. doi: 10.1016/j.injury.2024.111735. Epub 2024 Jul 25. PMID 39153311